CLINICAL TRIAL: NCT01473004
Title: An Open-Label, Single Institution, Phase II Study Using Radioactive Yttrium90 Microsphere (SIR-Sphere®) in Uveal Melanoma Patients With Hepatic Metastasis
Brief Title: SIR-Spheres® 90Y Microspheres Treatment of Uveal Melanoma Metastasized to Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10D.95; JT 2216 (Other: JeffTrial Number)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Stage IV Uveal Melanoma
Keywords: Sir-spheres; Liver Metastases; Selective internal radiation; Yttrium-90; Uveal; Melanoma; Ocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A: no prior intra-hepatic arterial treatment (Experimental): Patients with no prior intra-hepatic arterial treatment will be treated with intra-hepatic arterial infusion of Yttrium-90 radioactive microspheres (SIR-Spheres® microspheres). Sir-Spheres® Yttrium-90 microspheres given intra-hepatic; once for each lobe involved separated by 4 weeks.
  Interventions: Device: Sir-Spheres®
- Group B: one prior hepatic trans-arterial embolization treatment (Experimental): Patients with one prior hepatic trans-arterial embolization treatment will be treated with intra-hepatic arterial infusion of Yttrium-90 radioactive microspheres (SIR-Spheres® microspheres). Sir-Spheres® Yttrium-90 microspheres given intra-hepatic; once for each lobe involved separated by 4 weeks.
  Interventions: Device: Sir-Spheres®

INTERVENTIONS:
Device: Sir-Spheres® — Sir-Spheres® Yttrium-90 microspheres given intra-hepatic; once for each lobe involved separated by 4 weeks.

SUMMARY:
The purpose of this study is to determine whether radiation provided locally to the liver tumor vasculature environment will demonstrate a response of tumor decline. This radiation may cause the tumor cells to die.

This is a phase II clinical trial to investigate safety and efficacy of radioactive microsphere (SIR-Spheres® microspheres). Uveal melanoma patients with progressing hepatic metastases who received no more than one intra-hepatic arterial treatment will be enrolled. Patients will be first stratified into two groups: Group A, no prior intra-hepatic arterial treatment; Group B, one prior intra-hepatic arterial treatment).

DETAILED DESCRIPTION:
This is an open-label, uncontrolled single institution phase II study for metastatic uveal melanoma. Uveal melanoma patients who received one or less prior trans-arterial embolization treatment of hepatic metastasis are eligible. Patients will be stratified into two groups: Group A, no prior intra-hepatic arterial treatment, n=24; Group B, one prior hepatic trans-arterial embolization treatment, n=24. They will be treated with intra-hepatic arterial infusion of Yttrium-90 radioactive microspheres (SIR-Spheres® microspheres).

Within 4 weeks prior to radiosphere treatment, patients undergo the pre-assessment angiogram and technetium-99m-labelled macroaggregated albumin (99m Tc -MAA) nuclear scan to block the collateral flow to non-target organs and to calculate the shunting rate to the lung. Once patients meet the eligibility criteria of the study, the radiosphere treatment will be given. The Yttrium-90 radioactive microsphere treatment generally consists of two sequential uni-lobar treatments, approximately 4 weeks (3 to 5 weeks) apart. In selected patients, if clinically feasible, a biopsy of hepatic metastasis will be obtained prior to radiosphere treatment to investigate the correlation between efficacy of treatments and molecular characteristics of metastatic uveal melanoma.

The side effects of Yttrium-90 radioactive microspheres will be monitored every 2 weeks for one month following each treatment and then every month for three months after the last radiosphere treatment. The efficacy of radiosphere treatment will be evaluated every 3 months from the last treatment for 2 years until disease progression or death.

If patients experience grade 3 toxicity after the first treatment with Yttrium-90 radioactive microspheres, the second radiosphere treatment will be held until the resolution of toxicity to grade 1 or less or for a maximum of 6 weeks. The dose of the second radiosphere treatment will be decreased by 50% for liver-related grade 3 toxicity. A dose reduction will not be considered for grade 3 GI toxicity unless the next treatment is repeated to the same hepatic lobe. The study treatment will be discontinued for grade 4 toxicity or if patients do not recover from the grade 3 toxicity to at least a grade 1 within 6 weeks.

The study will require two years of accrual with an additional two years of follow-up for survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* must have diagnosis of metastatic melanoma liver disease by histological confirmation
* one measurable untreated or progressed liver lesion
* less than 50% liver involvement
* must have ECOG performance status of 0-1
* must have adequate renal and bone marrow function as: serum creatinine ≤ 2.0 mg/dl, granulocyte count ≥1000/mm3 and platelet count ≥100,000/mm3
* must have adequate liver function as: total bilirubin <1.6 mg/ml and albumin >3.0 g/dl

Exclusion Criteria:

* failure to meet any of the inclusion criteria
* solitary liver metastasis that is amenable to surgical removal
* previous treatment with isolated hepatic perfusion
* systemic chemotherapy within 2 weeks of study entry
* significant shunting to the lung (>20%) as identified on Technetium-99m-macro-aggregated albumin nuclear medicine break-through scan
* unsuccessful closure of collateral blood flows from the hepatic artery to non-targeted organs such as the GI tract
* symptomatic liver failure including ascites and hepatic encephalopathy
* metastasis outside of liver requiring systemic treatment within 3 months
* untreated brain metastasis
* main portal vein occlusion or inadequate collateral flow
* uncontrolled hypertension or congestive heart failure
* acute myocardial infarction within 6 months
* medical complications with implication of less than 6 month survival
* uncontrolled severe bleeding tendency or active GI bleed
* significant allergic reaction to iodinated contrast
* previous radiation that includes the liver in the main radiation field
* pregnant or breast-feeding women
* biliary obstruction, stent, or prior biliary surgery including sphincterotomy but excluding cholecystectomy
* children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takami Sato, MD, Principal Investigator — Thomas Jefferson University; Carin Gonsalves, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - No Prior Embolization: no prior intra-hepatic arterial treatment
- Group B - Prior Embolization: one prior hepatic trans-arterial embolization treatment
Period: Overall Study
Arm/Group | Group A - No Prior Embolization | Group B - Prior Embolization
Started | 24 | 24
Completed | 23 | 24
Not Completed | 1 | 0
Not completed — Incomplete Lobar Treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: no Prior Intra-hepatic Arterial Treatment | Group B: One Prior Hepatic Trans-arterial Embolization Treatment | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 77] | 59 [34 to 77] | 61 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 14 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate of Previously Treated and Naive Patients
Description: Evaluation of clinical benefit includes status of complete and partial response as well as stable disease
Time Frame: 3 months post final treatment, an average of 4 months
Population: Clinical response in the liver metastases will be evaluated 3 months after the last radiosphere treatment using CT scans or MRI of the abdomen. The same modality must be used for serial measurements of target lesions. The sum of the longest diameter (LD) of up to 5 target liver lesions will be used to determine response.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - No Prior Embolization | Group B - Prior Embolization
Number analyzed (Participants) | 24 | 24
Participants
  Complete Response | 0 | 0
  Partial Response | 7 | 6
  Stable Disease | 13 | 8
  Progressive Disease | 3 | 10
  Not Evaluated | 1 | 0

2. Primary Outcome: Number of Patients With Adverse Events
Description: Adverse events except for baseline symptoms will be collected from start of first treatment to 3 months post final treatment
Time Frame: 3 months post final treatment, an average of 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - No Prior Embolization | Group B - Prior Embolization
Number analyzed (Participants) | 24 | 24
Participants | 16 | 15

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is measured from the start of the treatment to patient death. Date and cause of death will be recorded. The cause of death will be categorized as either cancer-related or cancer-unrelated.
Time Frame: From date of first SIR-Spheres® administration until the date of death from any cause, assessed up to 6 years
Measure: Median (Full Range); unit: months
Arm/Group | Group A - No Prior Embolization | Group B - Prior Embolization
Number analyzed (Participants) | 24 | 24
months | 18.9 [6.5 to 66.9] | 19.1 [4.8 to 68.4]

4. Secondary Outcome: Progression Free Survival
Description: Period of time without progression of liver metastasis
Time Frame: 2 years post treatment, an average of 10 months
Measure: Median (Full Range); unit: months
Arm/Group | Group A - No Prior Embolization | Group B - Prior Embolization
Number analyzed (Participants) | 24 | 24
months | 8.1 [3.3 to 33.7] | 5.2 [2.9 to 22.0]

5. Secondary Outcome: Duration of Response
Time Frame: 2 years post treatment, an average of 10 months
Population: One participant from Group A was not evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A - No Prior Embolization | Group B - Prior Embolization
Number analyzed (Participants) | 23 | 24
months | 8.1 [6.4 to 11.8] | 5.2 [3.7 to 9.8]

ADVERSE EVENTS:
Time Frame: From first SIR-Spheres® administration through 3 months post-final treatment, up to 6 years.
Description: Adverse events were monitored and graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Events were recorded from the first administration of SIR-Spheres® Yttrium-90 microspheres through 3 months after the final treatment. Only treatment-emergent adverse events were included.
Arm/Group | Group A - No Prior Embolization | Group B - Prior Embolization
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 16/24 | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - No Prior Embolization (N=24) | Group B - Prior Embolization (N=24)
Abdominal Pain - Grade 1 (Gastrointestinal disorders) | 11 (11) | 3 (3)
Abdominal Pain - Grade 2 (Gastrointestinal disorders) | 3 (3) | 3 (3)
Allergy Antibiotic Eye Med - Grade 1 (Immune system disorders) | 1 (1) | 0 (0)
Anorexia - Grade 1 (Gastrointestinal disorders) | 5 (5) | 1 (1)
Anorexia - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthralgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Back Pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bladder - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Bladder - Grade 2 (Infections and infestations) | 0 (0) | 1 (1)
Bloating/Flatulence - Grade 1 (Gastrointestinal disorders) | 4 (4) | 3 (3)
Bloating/Flatulence - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blotchy Skin - Grade 1 (General disorders) | 3 (3) | 0 (0)
Bruising / hematoma groin - Grade 1 (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Bruise - Grade 1 (Vascular disorders) | 3 (3) | 2 (2)
Burning RUQ - Grade 1 (Gastrointestinal disorders) | 2 (2) | 0 (0)
Concentration Impairment - Grade 1 (Nervous system disorders) | 1 (1) | 0 (0)
Conjunctivitis - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diarrhea/ Constipation - Grade 1 (Gastrointestinal disorders) | 4 (4) | 6 (6)
Dizziness / Lightheadedness - Grade 1 (Nervous system disorders) | 0 (0) | 2 (2)
Dry Mouth - Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia - Grade 1 (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia - Grade 2 (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 3 (3) | 0 (0)
Edema - Grade 1 (General disorders) | 0 (0) | 3 (3)
Eye Pain - Grade 2 (Eye disorders) | 2 (2) | 0 (0)
Fatigue - Grade 1 (General disorders) | 16 (16) | 15 (15)
Fatigue - Grade 2 (General disorders) | 6 (6) | 2 (2)
Fever - Grade 1 (General disorders) | 0 (0) | 1 (1)
Flu / Sinusitis / Cold - Grade 1 (Infections and infestations) | 6 (6) | 6 (6)
Flu / Sinusitis / Cold - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Food Poisoning - Grade 2 (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fungal Skin Infection - Grade 1 (Infections and infestations) | 1 (1) | 0 (0)
Gastritis - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD/heartburn - Grade 1 (Gastrointestinal disorders) | 3 (3) | 4 (4)
GERD/heartburn - Grade 2 (Gastrointestinal disorders) | 1 (1) | 2 (2)
Headache - Grade 1 (Nervous system disorders) | 4 (4) | 2 (2)
Headache - Grade 2 (Nervous system disorders) | 1 (1) | 1 (1)
Hiccups - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperglycemia - Grade 1 (Gastrointestinal disorders) | 4 (4) | 9 (9)
Hyperglycemia - Grade 2 (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypersomnia - Grade 1 (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension/Atrial Fibrillation - Grade 1 (Cardiac disorders) | 3 (3) | 0 (0)
Hypotension/Atrial Fibrillation - Grade 2 (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Insomnia - Grade 1 (Psychiatric disorders) | 8 (8) | 2 (2)
Insomnia - Grade 2 (Psychiatric disorders) | 1 (1) | 0 (0)
Memory Impairment - Grade 1 (Nervous system disorders) | 0 (0) | 1 (1)
Mood Alterations - Grade 1 (Psychiatric disorders) | 2 (2) | 1 (1)
Mood Alterations - Grade 2 (Psychiatric disorders) | 1 (1) | 0 (0)
Nausea / Emesis - Grade 1 (Gastrointestinal disorders) | 11 (11) | 12 (12)
Nausea / Emesis - Grade 2 (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea / Emesis - Grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Night Sweats - Grade 1 (General disorders) | 0 (0) | 2 (2)
Pain - Grade 1 (General disorders) | 4 (4) | 9 (9)
Pain - Grade 2 (General disorders) | 0 (0) | 2 (2)
Pain - Grade 3 (General disorders) | 1 (1) | 0 (0)
Peripheral Neuropathy - Grade 1 (Nervous system disorders) | 1 (1) | 0 (0)
Pounding heartbeat/tightness - Grade 1 (Cardiac disorders) | 2 (2) | 0 (0)
Radiculitis - Grade 2 (Nervous system disorders) | 1 (1) | 0 (0)
Rib pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right leg/ Shoulder / Neck Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Right leg/ Shoulder / Neck Pain - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sedation - Grade 2 (Nervous system disorders) | 1 (1) | 0 (0)
Shortness of Breath - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore Throat - Grade 1 (General disorders) | 1 (1) | 0 (0)
Splenic Infarct - Grade 2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thromboembolic Event - Grade 3 (Vascular disorders) | 1 (1) | 0 (0)
Urinary Retention - Grade 2 (Renal and urinary disorders) | 1 (1) | 0 (0)
Varicose Veins - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)
Voice Change (transient) - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weight Loss - Grade 1 (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT01473004/Prot_SAP_000.pdf